CLINICAL TRIAL: NCT02056834
Title: Prospective, Multi-Center, Observational Study Evaluating the Augmentation With Calcium Phosphate Cement (chronOS Inject) for Bone Defect After Internal Fixation of Proximal Tibial Fractures
Brief Title: chronOS Inject in Proximal Tibial Fractures
Status: Completed | Type: Observational
Sponsor: Synthes GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: STU-BIO-T-XX-004-04
Record Dates: First submitted 2014-01-31; First posted 2014-02-06 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Closed Proximal Tibial Fracture Schatzker I - VI; Closed Proximal Tibial Fracture AO-OTA 41; Closed Proximal Tibial Fracture AO-OTA 42

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronOS Inject: Closed proximal tibial fractures of type Schatzker I - VI, AO-OTA 41, AO-OTA 42 with bone defect
  Interventions: Device: chronOS Inject

INTERVENTIONS:
Device: chronOS Inject — chronOS Inject is used as bone void filler in internal fixation of proximal tibial fractures

SUMMARY:
The primary objective of this study is to observe the safety, the radiological and clinical outcomes of chronOS Inject after having been used as bone void filler in internal fixation of proximal tibial fractures.

DETAILED DESCRIPTION:
The primary objective of this study was to observe the safety, the radiological and clinical outcomes of chronOS Inject after having been used as bone void filler in internal fixation of proximal tibial fractures. Secondary objectives were to assess the surgeon's satisfaction in using chronOS Inject and patient satisfaction post surgery.

The study was planned to be a multi-center, prospective, observational study. Patients with proximal tibial fractures of type Schatzker I - VI, AO-Müller-Orthopaedic Trauma Association (AO-OTA) 41, AO-OTA 42 with bone defect were assessed for eligibility to enter the study. Patients eligible for the study were followed over time to twelve months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with closed proximal tibial fractures defined by : Tibia plateau, Schatzker I - VI, AO-OTA 41, AO-OTA 42 with bone defect
* Skeletally mature adult 18 years or older, with close of growth plate at the time of surgery
* Psychosocially, mentally and physically able to fully comply with this protocol including adhering to scheduled visits, treatment plan, completing forms, and other study procedures
* Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Open fractures with severe soft tissue damage
* Proximal tibial fractures with tumor or osteomyelitis
* Any tibial anatomy or disease process that would interfere with deployment or performance of the device as defined by the surgeon
* Osteopenia or Osteoporosis: if dual energy x-ray absorptiometry (DEXA) is required, exclusion will be defined as a DEXA bone density measured T score <=-1.0
* Known history of Paget's disease, osteomalacia, or any other metabolic bone disease
* Morbid obesity defined as a body mass index >40 kg/m2 or weight more than 50 kg over ideal body weight
* Active malignancy. A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and there has been no clinical signs or symptoms of the malignancy >5 years
* Known or documented history of communicable disease, including AIDS and HIV
* Active Hepatitis (receiving medical treatment within two years)
* Active systemic or local infection
* Active rheumatoid arthritis, non-controlled diabetes mellitus, or any other medical condition(s) that would represent a significant increase in surgical risk or interfere with normal healing
* Current or recent history (within last 2 years) of substance abuse (e.g., recreational drugs, narcotics, or alcohol)
* Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for >1 month within last 12 months
* Pregnant or planning to become pregnant during study period
* Involved in study of another investigational product that may affect outcome
* History of psychosocial disorders that could prevent accurate completion of self reporting assessment scales
* Patients who are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proximal tibial fractures of type Schatzter I - VI, AO-OTA 41, AO-OTA 42 with bone defect are assessed for eligibility to enter the study. A computerized tomography is performed if necessary to confirm the fracture type and the amount of bone defect. Patients eligible for the study are followed over time to 12 months after surgery.
  A total of 30 patients who meet the inclusion/exclusion criteria are enrolled in the study, which is conducted at Kyungpook National University Hospital and Hanyang University Guri Hospital in the Republic of Korea.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Wug Oh, MD, Principal Investigator — Kyungpook National University Hospital; Kichul Park, MD, Principal Investigator — Hanyang University
Locations (2):
- South Korea (2):
  - Kyungpook National University Hospital, Daegu
  - Hanyang University Guri Hospital, Guri-si

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | chronOS Inject
Started | 36
6 Weeks | 34
6 Months | 31
Completed | 29
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | chronOS Inject
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (14.6)
Age, Customized [Number; unit: participants]
  Age group <=58 years | 19
  Age group >58 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 36
Smoking status [Number; unit: participants]
  Never | 23
  Former | 4
  Current | 9
Height [Mean (Standard Deviation); unit: cm] | 163.4 (8.99)
Weight [Mean (Standard Deviation); unit: kg] | 62.6 (12.15)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 23.3 (3.67)
Exercise per week [Number; unit: participants]
  Never | 9
  1-2 times per week | 21
  3-4 times per week | 5
  5 or more times per week | 1
Health status [Number; unit: participants]
  Excellent | 4
  Good | 28
  Fair | 3
  Poor | 0
  Missing | 1
Occupation [Number; unit: participants]
  Student | 3
  Office worker | 5
  Home worker | 7
  Retired | 6
  Light industrial or light industrial labour | 6
  Moderate industrial or moderate physical labour | 5
  Other | 4
Preoperative medical condition [Number; unit: participants]
  None | 22
  Any | 14
Preoperative medical conditions (description) [Number; unit: participants] — Subjects can have more than one medical condition.
  participants
    Adiposity | 1
    Allergies | 0
    Cancer | 0
    Cardiac | 4
    Congenital | 0
    Dermatological | 1
    Endocrine | 4
    Hematologic | 0
    Implants/Prosthesis | 0
    Infection | 0
    Musculoskeletal including fractures | 0
    Neurologic | 1
    Psychiatric | 0
    Respiratory | 2
    Urogenital | 0
    Vascular | 3
    Other | 3
Accident type [Number; unit: participants] — Patients can have more than one accident type.
  participants
    Sport | 1
    Low energy | 1
    High energy | 23
    Direct blow | 9
    Fall from height | 3
    Simple fall | 3
    Motorcycle accident | 4
    Pedestrian in traffic accident | 11
    Car occupant in traffic accident | 7
    Other | 2
Fracture type [Number; unit: participants] — Patients can have more than one fracture type.
  participants
    Schatzker Type I (lateral split) | 1
    Schatzker Type II (split with depression) | 14
    Schatzker Type III (pure lateral depression) | 0
    Schatzker Type IV (pure medial depression) | 2
    Schatzker Type V (bicondylar) | 6
    Schatzker Type VI (split extends to metadiaphysis) | 10
    AO-OTA 41 (proximal tibia fracture) | 29
    AO-OTA 42 (diaphyseal tibia fracture) | 0

OUTCOME MEASURES:

1. Primary Outcome: Fracture Union
Description: Fracture union (complete bone healing) was assessed by the investigators based on anteroposterior and lateral X-rays
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants
  Union | 27
  Non-union | 2

2. Primary Outcome: Articular Subsidence
Description: Evidence of articular subsidence (collapse of surface pertaining to the joint) of ≥2 mm was assessed by the investigators
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants
  Absent | 28
  Present | 1

3. Secondary Outcome: Absorption Rate of Calcium Phosphate Cement
Description: Absorption of calcium phosphate cement over time was calculated from X-rays with the INFINITT program.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of absorption at 12 months
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
percentage of absorption at 12 months | 0.64 (0.115)

4. Secondary Outcome: Patients Who Reached Full Weight Bearing
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants | 29

5. Secondary Outcome: Total Range of Motion
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants
  At least 140 degree | 17
  At least 120 degree | 11
  At least 90 degree | 1
  At least 60 degree | 0
  At least 30 degree | 0

6. Secondary Outcome: Anatomical Gradings Assessed Radiographically
Description: The following was assessed:
  * depression of knee joint: presence or absence
  * condylar widening (enlargement of the knee joint): presence or absence
  * angulation; valgus/varus (abnormal outward/inward turning of the knee): presence or absence
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants
  Absence of depression | 28
  Absence of condylar widening | 28
  Absence of angulation | 29

7. Secondary Outcome: Patient's Satisfaction
Description: Satisfaction with treatment was assessed by the subjects, where subjects indicated their satisfaction with treatment on a 100-mm visual analog scale. A score of zero indicated no satisfaction, while a score of 100 indicated completely satisfied.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
units on a scale | 80.52 (16.02)

8. Secondary Outcome: Surgeon's Satisfaction With the Product
Description: Satisfaction with product was assessed by the surgeon post-operatively, where surgeons indicated their satisfaction with treatment on a 100-mm visual analog scale. A score of zero indicated absolutely unacceptable, while a score of 100 indicated very satisfying.
Time Frame: Post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Inject
Number analyzed (Participants) | 36
units on a scale
  Mixing ability | 87.3 (6.16)
  Injecting ability | 87 (6.31)
  Application time | 87 (6.31)
  Moldability | 81.7 (9.59)
  Setting time | 77.1 (13.54)
  Rate of chronOS over bone graft | 68.6 (28.39)

9. Secondary Outcome: Extension Ability and Stability
Description: The following was assessed:
  * extension ability of the knee
  * stability of the knee in extension
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants
  Normal extension ability | 26
  0-10 degree extension ability | 3
  Normal extension stability | 28
  Abnormal extension stability | 1

10. Secondary Outcome: Peri-operative Complications
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 36
participants
  Microscopic or radiologic cement leakage during OP | 0
  Breakage of fixing device post-OP | 0
  Re-OP during hospital stay | 0
  Suffer from surgical wound complication post-OP | 0

11. Secondary Outcome: SF-12 Short Form Health Survey Physical Composite Score (PCS)
Description: The SF-12 short form health survey was self-administered to subjects preoperatively and all follow up visits. This health survey comprises 12 questions related to health and wellbeing over the prior four weeks. The responses to these 12 questions are entered into a standardized algorithm to provide summaries of physical and mental health (i.e., physical composite score [PCS] and mental composite score [MCS]). The summary scores are standardized and normalized such that a score of 50 for either the PCS or MCS corresponds to that of an average, healthy person. A score lower than 50 indicates poorer physical and mental health compared to an average, healthy person.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
units on a scale
  Score at baseline | 37.02 (9.616)
  Score at 12 months | 42.43 (4.589)
Statistical Analysis 1: Comparison: chronOS Inject; Paired T-Test p-value tests the significance of the percent change from baseline within each treatment group; Test type: Superiority or Other; p = 0.0166, t-test, 2 sided

12. Secondary Outcome: SF-12 Short Form Health Survey Mental Composite Score (MCS)
Description: The SF-12 short form health survey was self-administered to subjects preoperatively and at follow up visits. This health survey comprises 12 questions related to health and wellbeing over the prior four weeks. The responses to these 12 questions are entered into a standardized algorithm to provide summaries of physical and mental health (i.e., physical composite score [PCS] and mental composite score [MCS]). The summary scores are standardized and normalized such that a score of 50 for either the PCS or MCS corresponds to that of an average, healthy person. A score lower than 50 indicates poorer physical and mental health compared to an average, healthy person.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
units on a scale
  Score at baseline | 46.3 (9.707)
  Score at 12 months | 46.45 (7.145)
Statistical Analysis 1: Comparison: chronOS Inject; Paired T-Test p-value tests the significance of the percent change from baseline within each treatment group; Test type: Superiority or Other; p = 0.3785, t-test, 2 sided

13. Secondary Outcome: VAS Leg Pain Intensity
Description: The subjects completed questionnaires assessing the intensity and frequency of pain experienced in the leg at the baseline visit and postoperatively. Pain intensity was rated on a 100-mm visual analog scale where zero indicated no pain at all, and 100 represented the worst possible pain.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
units on a scale
  Score at baseline | 61.19 (32.714)
  Score at 12 months | 17 (18.592)
Statistical Analysis 1: Comparison: chronOS Inject; Paired T-Test p-value tests the significance of the change from baseline within treatment group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

14. Secondary Outcome: VAS Leg Pain Frequency
Description: The subjects completed questionnaires assessing the intensity and frequency of pain experienced in the leg at the baseline visit and postoperatively. Pain frequency was rated on a 100-mm visual analog scale where zero indicated no pain at all and 100 represented pain always.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
units on a scale
  Score at baseline | 57.28 (33.505)
  Score at 12 months | 20.52 (20.051)
Statistical Analysis 1: Comparison: chronOS Inject; Paired T-Test p-value tests the significance of the change from baseline within treatment group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

15. Secondary Outcome: Lysholm Knee Scale
Description: The Lysholm knee scale is a condition-specific outcome measure that was originally designed to assess ligament injuries of the knee. The survey was administered to subject at follow-up visits and comprises 8 subscales related to limp, support, stair climbing, squatting, walking, running and jumping as well as a question related to the atrophy of the thigh. The responses to these 8 questions are graded to provide a maximum result of 100 points.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | chronOS Inject
Number analyzed (Participants) | 29
participants
  Excellent (95-100) | 14
  Good (84-94) | 11
  Fair (65-83) | 3
  Poor (<65) | 1

16. Primary Outcome: Mean Time to Union
Description: Mean time to union was calculated based on the Kaplan-Meier estimator of the survivorship function
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | chronOS Inject
Number analyzed (Participants) | 34
months | 7.5 (0.441)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from treatment (implantation of the device) through the end of the follow-up period at 12 months.
Arm/Group | chronOS Inject
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 9/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | chronOS Inject (N=36)
Non-union of lateral tibial condyle (Musculoskeletal and connective tissue disorders) | 1 — Operative action taken (autogenous cancellous bone graft)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | chronOS Inject (N=36)
K-wire irritation (Skin and subcutaneous tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Volar mass on finger (MP joint) (Musculoskeletal and connective tissue disorders) | 1 (1)
Articular subsidence, loss of reduction and depression of lateral condyle of the tibia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1) — Drug treatment with Synerjet, Stillen and O Grand on April 8, 2011 (at 6 Months follow-up)
Cartilage damage at the initial injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Posterior neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-union of lateral tibial condyle (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less